CLINICAL TRIAL: NCT01679353
Title: Comparison of Analgesic Effect of Magnesium Added to Ropivacaine and Ropivacaine Alone in Caudal Analgesia on Postoperative Pain Control in Pediatric Patients Undergoing Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2012-0278
Record Dates: First submitted 2012-08-27; First posted 2012-09-06 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia, caudal analgesia, magnesium
MeSH Terms: conditions — Hernia, Inguinal | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo group (Placebo Comparator): normal saline 0.5ml
  Interventions: Drug: normal saline 0.5ml
- magnesum group (Experimental): After inhalation induction of general anesthesia, caudal block was applied. Patients were randomly assigned in two groups. Normal saline 0.5mL added to ropivacaine 0.15% 1.0 ml/kg was administered to Group R , Magnesium 50mg (Magnesium 10% 0.5mL)added to ropivacaine 0.15% 1.0ml/kg to Group MR.
  Interventions: Drug: caudal block

INTERVENTIONS:
Drug: caudal block — After inhalation induction of general anesthesia, caudal block was applied. Patients were randomly assigned in two groups. Normal saline 0.5mL added to ropivacaine 0.15% 1.0 ml/kg was administered to Group R , Magnesium 50mg (Magnesium 10% 0.5mL)added to ropivacaine 0.15% 1.0ml/kg to Group MR.
  Arms: magnesum group
Drug: normal saline 0.5ml
  Arms: placebo group

SUMMARY:
A caudal anesthesia is one of the most commonly used technique providing intra and postoperative analgesia in pediatric low abdominal surgery. The practice of adding adjunct analgesic drugs to local anesthetics for caudal block is common. The most commonly used drugs are opioids, clonidine, and ketamine. However, their use has been limited by adverse effects in children.

Recently, the importance of magnesium in analgesic effects has been increased. Magnesium is the fourth most abundant cation in the body. It has antinociceptive effects in human and these effects are primarily based on the regulation of calcium influx into the cell. Magnesium is a physiological calcium antagonist and blocks N-methyl-D-aspartate (NMDA) receptor and such NMDA antagonism prevents the central sensitization from nociceptive stimulation. Many study suggested that epidurally administered magnesium could reduce the postoperative pain in adults. But few studies are available about the use of magnesium in pediatrics.

The investigators performed prospective randomized double-blind study to examine the analgesic effect of magnesium added to ropivacaine and ropivacaine alone in caudal analgesia on postoperative pain control in pediatric patients undergoing inguinal hernia repair.

80 children (aged 2- 6 yr) undergoing inguinal hernia repair were included in this prospective, randomized, double-blinded study. After inhalation induction of general anesthesia, caudal block was applied. Patients were randomly assigned in two groups. Normal saline 0.5mL added to ropivacaine 0.15% 1.0 ml/kg was administered to Group R , Magnesium 50mg (Magnesium 10% 0.5mL)added to ropivacaine 0.15% 1.0ml/kg to Group MR. Postoperative pain was recorded at 30min and 1,2,3 h by using Hospital of Eastern Ontario Pain Scale (CHEOPS, 0-10) and Faces Legs Activity Cry Consolability tool (FLACC, 0-10). Participants will be followed for the duration of hospital stay, an expected average of 3 hours.

After discharge, rescue analgesic consumption, pain scores (Parents Postoperative Pain Measurement, PPPM), and adverse effects were evaluated for 48h.

The time to first supplemental oral analgesic medication demand was defined as the time from the end of surgery to the first registration of a PPPM( 0 - 15) ≥ 6 by parent's observation. 48 hours after surgery, reports of delayed side effects and demands for rescue analgesics from the child were gathered from parents via a telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I-II,
* children aged 2 to 6 yr
* weight under 20kg
* undergoing inguinal hernia repair

Exclusion Criteria:

* Hypersensitivity fo any local anesthetics,
* bleeding diathesis, infections at puncture sites,
* pre-existing neurological disease,
* patients taking Calcium channel block,
* patients taking opioid

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The number of children who required analgesics | at 24 and 48 hours after surgery
  Primary outcome is defined as the number of patients who required analgesics after discharge. Postoperative pain at home is assessed by parent using the PPPM scale that consists of 15 questions requiring a "yes" or "no" answer (yes = 1 point and no = 0 point). A PPPM score ≥ 6 by parent's observation is considered to represent clinically significant pain, requiring analgesics.
  The PPPM is a 15-item observational checklist measure of pain intensity that was designed to be used by parents to support research and clinical postoperative care for children at home.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Farouk S. Pre-incisional epidural magnesium provides pre-emptive and preventive analgesia in patients undergoing abdominal hysterectomy. Br J Anaesth. 2008 Nov;101(5):694-9. doi: 10.1093/bja/aen274. Epub 2008 Sep 26. PMID 18820247